CLINICAL TRIAL: NCT03059888
Title: Pilot Trial of Orencia in Myasthenia Gravis Patients Inadequately Responsive to Conventional Immunotherapy
Brief Title: Trial of Orencia in Patients With Myasthenia Gravis
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Mutual decision of sponsor and investigator due to logistical challenges
Sponsor: Johns Hopkins University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00100059
Record Dates: First submitted 2017-02-17; First posted 2017-02-23 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Abatacept (Experimental): 125mg abatacept in 1ml solution administered once per week by subcutaneous injection
  Interventions: Drug: Abatacept Injection

INTERVENTIONS:
Drug: Abatacept Injection — Subcutaneous administration of abatacept
  Other Names: Orencia

SUMMARY:
This pilot research study is being done to see if the drug abatacept (Orencia ®) will be helpful in treating patients with myasthenia gravis (MG) who do not respond satisfactorily to other drugs that are used to suppress the immune system. Abatacept has been successful in treating experimental MG in laboratory animals, and this study is to determine its effectiveness in patients with MG.

ELIGIBILITY:
Inclusion Criteria:

* Able to comprehend and willing to sign an Informed Consent Form (ICF)
* Male or female 16 to 85 years of age
* Diagnosis of DEFINITE Myasthenia Gravis
* History of inadequate response to conventional MG treatment
* Clinical laboratory findings within the normal range or, if outside the normal range, deemed not clinically significant by the Investigator
* Female patients of childbearing potential who are not be breastfeeding, have a negative pregnancy test, have no intention to become pregnant during the course of the study, and are using contraceptive drugs or devices to prevent pregnancy during their participation in the study
* Willing to cooperate with study requirements, including visits to the study site every 2 months.

Exclusion Criteria:

* Subject's MG is responding adequately to conventional immunosuppressive treatment
* Subject has had no previous trial of other immunosuppressive agents
* Subject has a history of Chronic Obstructive Pulmonary Disease (COPD)
* Subject is impaired, incapacitated or incapable of completing study-related assessments
* Subject has the presence at screening of any severe, progressive or uncontrolled renal, hepatic, hematologic, gastrointestinal, pulmonary, cardiac, neurologic or cerebral disease, whether or not related to MG that, in the opinion of the Investigator, might place the subject at unacceptable risk for participation in the study.
* Female subject has a history of breast cancer screening that is suspicious for malignancy and in whom the possibility of malignancy cannot be reasonably excluded by additional clinical, laboratory or other diagnostic evaluations
* Subject has a history of cancer in the last 5 years, other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ
* Subject currently abuses drugs or alcohol
* Subject has evidence of active or latent bacterial or viral infections, including positive infectious disease laboratory test result (Hepatitis B, Hepatitis C or HIV)
* Subject has history of herpes zoster or cytomegalovirus (CMV) infection that resolved less than 2 months prior to screening visit
* Subject has received any live vaccine within 3 months of screening
* Subject has a history of serious bacterial infection within in the last 3 months, unless treated and resolved with antibiotics; or, any chronic bacterial infection
* Subject is at risk for tuberculosis
* Subject has any of the following laboratory values: Hemoglobin < 8.5 g/dL; White Blood Cells (WBC) < 3000 mm3; Platelets < 100,000 mm3; Serum creatinine > 2x upper limit of normal (ULN); Serum Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) > 2x ULN
* Subject is unable or unwilling to maintain weekly injection schedule
* Subject has undergone a change in immunosuppressive medications within the last three months prior to enrollment.
* Subject has neurological impairment due to a condition other than MG, including history of transient ischemic attack within the past year
* Subject has taken any investigational study drug within 28 days or five half-lives of the prior agent, whichever is greater, prior to dosing
* Subject has had previous exposure to Orencia (abatacept)
* Subject is a prisoner or is involuntarily incarcerated
* Subject is compulsorily detained for treatment of either psychiatric or physical illness
* Subject is judged to be actively suicidal or a suicide risk by the Investigator

Ages: 16 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2017-04-12 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2019-07-15 (Actual)

PRIMARY OUTCOMES:
Subjective Composite Score of Myasthenia Gravis (MG) Severity | 12 months
  The "Subjective Score of MG Severity" is a composite score of subjective measurements of MG severity as designed by Dr. Daniel Drachman. The investigator will rate each subjective measure on a scale of 0 (no impairment) to 3 (severe impairment). The composite score of these measurements determined at baseline and at two-month increments through 12 months. The domains that make up the subjective score are: Diplopia, Ptosis, Arm strength, Leg strength, Speech, Voice, Chewing, Swallowing, Respiration, and General Health Status. The change in the composite subjective score at 12 months as compared to baseline is one of the primary outcomes. Patients that show an improvement in MG symptoms should have a lower score at 12 months as compared to baseline.
Objective Composite Score of Myasthenia Gravis (MG) Severity | 12 months
  The "Objective Score of MG Severity" is a composite score of subjective measurements of MG severity as designed by Dr. Daniel Drachman. The investigator will score each objective measure on a scale of 0 (no impairment) to 3 (severe impairment). The composite score of these measurements determined at baseline and at two-month increments through 12 months. The domains that make up the objective score are: Diplopia, Ptosis, Arm abduction, Gait, Orbicularis Oculi, Orbicularis Oris, Tongue, Slurp Test. The change in the composite objective score at 12 months as compared to baseline is one of the primary outcomes. Patients that show an improvement in MG symptoms should have a lower score at 12 months as compared to baseline.
Muscle Strength (Dynamometry) | 12 months
  Muscle strength in 11 muscle groups will be measured by hand-held dynamometry at baseline and at two-month increments through 12 months. The change in muscle strength (in pounds) at 12 months as compared to baseline is one of the primary outcomes. Patients that show an improvement in MG symptoms should show increased muscle strength at 12 months as compared to baseline.

SECONDARY OUTCOMES:
Myasthenia Gravis Composite Score (MGC) | 12 months
  The Myasthenia Gravis Composite (MGC) scale consists of test items that measure symptoms and signs of MG, with weighted response options. The domains included in the MGC are: Ptosis, Double vision, Eye closure, Talking, Chewing, Swallowing, Breathing, Neck strength, Shoulder abduction and Hip flexion. Each domain is rated by the Investigator on a weighted scale between 0 (no impairment) and 6 (severe impairment). Patients that show an improvement in MG symptoms should have a lower score at 12 months as compared to baseline.
Myasthenia Gravis Quality of Life-15 (MG QOL15) Score | 12 months
  The MG-QOL15 is a brief survey, completed by the patient, that is designed to assess some aspects of "quality of life" related to myasthenia gravis. Patients are given 15 statements that relate to their quality of life and are asked to chose how often that statement applies to them (Not At All, A Little Bit, Some-what, Quite A Bit, Very Much). Their answers are assigned a score from 0 (not at all) to 4 (Very Much). Patients that show an improvement in quality of life as related to their MG symptoms should have a lower score at 12 months as compared to baseline.
Acetylcholine Receptor (AChR) or Muscle-Specific Kinase (MuSK) Antibody Concentrations | 12 months
  For patients with positive AChR or MuSK antibody tests, the change in antibody concentration will be a secondary outcome. Patients with MG will only be positive for one of these antibodies. Improvement is often seen with reduction in titer of > 50%, therefore patients that show an improvement in MG symptoms should show a reduction in antibody levels at 12 months as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Drachman, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No